CLINICAL TRIAL: NCT06507670
Title: Point of Care Ultrasound for the Detection of Esophageal Food Bolus
Status: Recruiting | Type: Observational
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Brent Becker, Research Director - Department of Emergency Medicine, WellSpan Health
Other Study IDs: 2207289
Record Dates: First submitted 2024-07-05; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Foreign Body; Esophageal Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Esophageal foreign body/impaction (suspected)
  Interventions: Diagnostic Test: Point of care ultrasound
- Control (No symptoms of esophageal foreign body/impaction)
  Interventions: Diagnostic Test: Point of care ultrasound

INTERVENTIONS:
Diagnostic Test: Point of care ultrasound — Point of care medical ultrasound machines will be used to sonographically visualize the esophagus and following sonographic data will be collected:
  * Presence/absence of suspected foreign body
  * Sonographic esophageal measurements (diameters, area)
  * Other relevant secondary sonographic findings

SUMMARY:
This will be a prospective, observational, case-control study of adult patients presenting to the WellSpan York Hospital Emergency Department (YHED) with signs and symptoms of esophageal food or foreign body impaction. Point of care ultrasound (POCUS) will then be performed by a trained emergency physician to collect ultrasound data, including the presence or absence of direct visualization food bolus/foreign body, as well as secondary markers of dilatation, such as maximal esophageal area. Investigators will also enroll an age/sex-matched control group of asymptomatic individuals to establish baseline esophageal measurements.

Patients will otherwise receive medical treatment per standard of care. Subsequent interventions will also be documented, including glucagon, carbonated beverages, and esophagogastroduodenoscopy (EGD). If patients remain in the ED and improve without need for EGD they will undergo repeat ultrasound. Chart review at 1 month will be performed to establish results of EGD including improvement, recurrence, or presence of pathologic abnormalities. The investigators aim to establish normal and abnormal parameters to aid in the diagnosis of esophageal food impactions to predict need for definitive EGD management.

ELIGIBILITY:
Eligibility (CASES)

* Inclusion criteria:

  1. Age ≥18 years
  2. Signs and symptoms of esophageal food bolus or foreign body
* Exclusion criteria:

  1. Prior esophageal surgery
  2. History of head/neck cancer
  3. Incarcerated individuals
  4. Individuals unable to provide consent
  5. Clinical instability or airway compromise

Eligibility (CONTROLS)

* Inclusion criteria:

  1. Age ≥18 years
  2. NO signs or symptoms of esophageal food bolus or foreign body
  3. Age/Sex match to previously enrolled case subject
* Exclusion criteria:

  1. Prior esophageal surgery/dilation/pathology
  2. History of head/neck cancer
  3. Incarcerated individuals
  4. Individuals unable to provide consent
  5. Clinical instability or airway compromise
  6. Presentation involving any of the following symptoms:
* Nausea/vomiting
* Diarrhea
* Abdominal pain
* Chest pain
* Shortness of breath
* Dysphagia/odynophagia
* Cough

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This will be a case-control study of adult patients presenting to the WellSpan York Hospital Emergency Department (YHED) with signs and symptoms of esophageal food or foreign body impaction. We will also enroll an age/sex-matched control group of asymptomatic individuals to establish baseline esophageal measurements.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of esophageal foreign body/food impaction | Within 48 hours of index visit (Emergency department arrival to emergency department or hospital discharge)
  Presence of absence of esophageal foreign body/food impaction on esophagogastroduodenoscopy

SECONDARY OUTCOMES:
Number/proportion of subjects experiencing resolution of symptoms with standard medical therapies | Within 48 hours of index visit (Emergency department arrival to emergency department or hospital discharge)
  Number/proportion of subjects experiencing resolution of symptoms with standard medical therapies, including glucagon and carbonated beverages
Number/proportion of subjects requiring endoscopic intervention | Within 48 hours of index visit (Emergency department arrival to emergency department or hospital discharge)
  Number/proportion of subjects needing interventional procedures during esophagogastroduodenoscopy due to esophageal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- WellSpan Health York Hospital, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No